CLINICAL TRIAL: NCT06320873
Title: The Effect of Pulmonary Functions and Respiratory Muscle Strength on Sports Performance in Elite Archers
Brief Title: The Effect of Respiratory on Sports Performance in Archers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: zselcuk1
Record Dates: First submitted 2024-02-15; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Sports Physical Therapy
MeSH Terms: interventions — Employee Performance Appraisal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Results of sports performance parameters values in archers (Other): Sociodemographic and physical characteristics, Pulmonary function test (PFT), respiratory muscle strength, shooting performance test, Moberg-pickup collection test, Nelson hand reaction test, and Fatigue Severity Scale (FSS)
  Interventions: Other: archery respiratory parameters

INTERVENTIONS:
Other: archery respiratory parameters — Evaluation of respiratory functions, respiratory muscle strength and shooting performance in archers
  Other Names: performance evaluation

SUMMARY:
Purpose: The physical, physiological, and functional characteristics of archers affect target shooting performance. In our study, we aimed to examine the effect of pulmonary functions and respiratory muscle strength on sports performance in archers.

Methods: Our study included 46 (27 female, 19 male) professional archers registered in archery sports clubs. Sociodemographic and physical characteristics were recorded. Pulmonary function test (PFT), respiratory muscle strength, shooting performance test, Moberg-pickup collection test, Nelson hand reaction test, and Fatigue Severity Scale (FSS) were applied to all participants.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-30 years old,
* Professional archers.

Exclusion Criteria:

* Participants who had COVID-19 (Coronavirus Disease) in the last 2 months,
* Musculoskeletal disorders,
* Orthopedic surgery,
* Smoking history,
* Neurologic and pulmonary diseases.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
FEV1 (liter) | at the enrollment
  This is the amount of air with pulmonary function test that the patient can force out of their lungs in one second.
FEV1 (%-percentage) | at the enrollment
  This is the percentage of air with pulmonary function test that the patient can force out of their lungs in one second.
FVC (liter) | at the enrollment
  This is the greatest total amount of air patient can forcefully breathe out after breathing in as deeply as possible.
FVC (%-percentage) | 7 months
  This is the percentage of air patient can forcefully breathe out after breathing in as deeply as possible.
FEV1/FVC (percentage) | at the enrollment
  The FEV1/FVC ratio is a number that represents the percentage of patient lung capacity patient is able to exhale in one second.
Inspiratory muscle test | at the enrollment
  Maximal inspiratory pressure (MIP) is going to measured using a mouth pressure meter (MicroRPM; MicroMedical, UK) according to the guideline of ATS and European Respiratory Society (ERS).
Expiratory muscle test | at the enrollment
  Maximal expiratory pressure (MEP) is going to measured using a mouth pressure meter (MicroRPM; MicroMedical, UK) according to the guideline of ATS and European Respiratory Society (ERS).
Shooting performance | at the enrollment
  The high shooting score indicates high arrow shooting performance.
Nelson Hand Reaction Test | at the enrollment
  The average value when the participants catch the ruler for three attempts
Moberg-pickup collection test | at the enrollment
  Assess manual dexterity and function by measuring the time it takes to pick up twelve different small objects (screws, paper clips, rings, safety pins, small nuts, coins, and wrenches)
The Fatigue Severity Scale (FSS) | at the enrollment
  Assess fatigue severity with 9-item self reporting scale

CONTACTS AND LOCATIONS:
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No